CLINICAL TRIAL: NCT06582992
Title: EPIGENETIC-SENSITIVE BIOMARKERS OF INFLAMMAGING FROM HEALTHY TO HEART FAILURE DISEASE
Brief Title: DNA Methylation Trajectories in Aging
Acronym: EPI-GERAS
Status: Not yet recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Giuditta Benincasa, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: Aging Well in an Aging Society
Record Dates: First submitted 2024-08-31; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Aging
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Isolation of circulating T lymphocytes and DNA extraction; isolation of plasma and protein detection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Young healthy subjects: This cohort is characterized by 50 healthy subjects aged < 40 years (blood donor volonteers)
  Interventions: Other: RRBS
- Aged healthy subjects: This cohort is characterized by 50 healthy subjects aged > 60-65 years (blood donor volonteers) without signs and symptoms of heart failure
  Interventions: Other: RRBS
- Patients with heart failure: This cohort is characterized by 50 subjects aged > 60-65 years with signs and symptoms of heart failure with preserved ejection fraction
  Interventions: Other: RRBS

INTERVENTIONS:
Other: RRBS — Measure of genomic regions with differentially methylated profiles and differentially expressed protein
  Other Names: O-Link Targeted Proteomics

SUMMARY:
The goal of this observational study is to profile changes in DNA methylation of circulating CD4+ T and CD8+ T cells from healthy young to aged with diagnosis of HFpEF, a particular phenotype of HF which is highly prevalent in aging.

The main question it aims to answer is:

-Do DNA methylation biomarkers help us to understand the role of inflammation in HFpEF during aging?

Our goal is to provide a simple large-scale panel of epigenetic-sensitive biomarkers useful in aged patients with HF in the early natural history of the disease (HFpEF).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged between 18 and 40 years
* Aged subjects (≥65) without signs and symptoms of heart failure
* Aged subjects (≥65) with diagnosis of heart failure with preserved ejection fraction (EF major than 50%)

Exclusion Criteria:

* Heart failure with reduced ejection fraction (EF minor than 40%)
* Heart failure with mildly reduced EF (HFmrEF) (EF 41-49%)
* History or diagnosis of cancer and inflammatory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 150 subjects will be enrolled; n=50 healthy young, n=50 aged (≥65) without signs and symptoms of heart failure, and n=50 aged (≥65) with diagnosis of HFpEF will be enrolled at Trasfusion Medicine and Cardiology Departments of University of Campania Luigi Vanvitelli; Each group will be matched for sex (25 M and 25 F), smoker habits, and comorbidities. Demographic and clinical characteristics will be collected both from patients and healthy subjects at baseline. For HFpEF patients, echocardiographic parameters will be reported based on the echocardiogram acquired at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of differentially methylated positions and regions as assessed by RRBS | 6 months
  We will identify a panel of positions and regions of the genome which are differentially methylated using as measure diff.meth more than or minor than 2 and p minor than 0.05

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania Luigi Vanvitelli, Naples, No States Available, Italy

IPD SHARING:
Plan to Share IPD: No
Not required